CLINICAL TRIAL: NCT05845177
Title: Incidence of Persistent Pain After Total Hip Arthroplasty: A Nationwide Cross-sectional Survey Study
Brief Title: Persistent Pain After Hip Replacement
Status: Completed | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Jens Laigaard, Principal investigator, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: P-2022-933
Record Dates: First submitted 2023-04-06; First posted 2023-05-06 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Persistent Postsurgical Pain; Arthritis Hip; Neuropathic Pain; Opioid Use
MeSH Terms: conditions — Pain, Postoperative; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Primary Total Hip Arthroplasty — All patients surveyed have undergone primary total hip arthroplasty approximately 1 year prior to survey distribution
  Other Names: Primary Total Hip Replacement

SUMMARY:
This study is a nationwide cross-sectional survey on pain and satisfaction after total hip arthroplasty (THA). Please find the full protocol uploaded on ClinicalTrials.gov

DETAILED DESCRIPTION:
The study is registered at the Capitol region of Denmark's regional research listing (Pactius) with identifier P-2022-933, approved 23 December 2022. The resulting paper will be reported according to the CROSS checklist for standardised reporting of survey studies. Wherever needed, a trained linguist translated questions from English to Danish and vice versa. The Danish and an English version of the questionnaire will be available in the final publication.

* Study design: This study is a nationwide cross-sectional survey.
* Patient involvement: A panel of patients helped develop the questionnaire, i.e. testing and selecting the questions.
* Questionnaire: The questionnaire is composed of 22 questions (please see the uploaded protocol), however patients answering "No" to question 3 skips questions 4-17 concerning pain in the operated hip. Only question 3, 4, 20, and 21 are mandatory as to avoid non-respondents. The full questionnaire translated to English can be found in the supplementary material in the protocol. Contact information for the first author (JL) is supplied in the contact letter in case the patients have difficulties with filling in the questionnaire, have questions, or believe they have been selected mistakenly. Similar or identical questions to those in a survey published in 2006 to increase the ability to compare results (i.e., questions 3-5, 8, 10 and 13)
* Sample characteristics: Eligible patients are all adult (18 years or older) patients operated with primary THA for osteoarthritis between 1 March and May 31, 2022. Legally incompetent citizens, i.e., persons with a legal guardian, will not be asked to participate. Patients will be identified from the Danish National Patient Register through the Danish Health Data Authority (SKS-code DM16 [hip osteoarthritis] + KNFB [Primary Total Hip Arthroplasty]). Baseline data of respondents and non-respondents are gathered from the Danish Hip Arthroplasty Register. To evaluate the generalisability of the study, respondents' baseline data will be compared to the non-respondents baseline data in the paper's Table 1.
* Sample size calculation: With an estimated 12% incidence of the primary outcome (patients with moderate or severe pain at rest and/or while walking) and a 70% response rate, 2577 patients are needed to yield a 95% confidence interval of 3 percentage points (10.5-13.5). This level of certainty is appropriate because differences less than this, may be hard to interpret by clinicians and patients. Sampling patients that were operated during 3 months outside holiday season should yield approximately this number of identified patients.
* Ethical considerations: This study was approved by the local institutional review board and contact information are provided by the Danish Health Data Authority. Telephone numbers for non-respondents are found by searching the CPR number in the electronic patient files, but without accessing the patients' health data. According to Danish legislation, approval from the national ethics committee is neither required nor possible to obtain for survey studies (see attached 'exempt from notification' letter from the Danish national ethics committee).

ELIGIBILITY:
Inclusion Criteria:

* Patients operated with primary THA for osteoarthritis 12-15 months before survey distribution

Exclusion Criteria:

* Legally incompetent citizens, i.e., persons with a legal guardian, will not be asked to participate.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are identifed from the Danish National Patient Register through the Danish Health Data Authority (SKS-code DM16 [hip osteoarthritis] + KNFB [Primary Total Hip Arthroplasty]). Baseline data of respondents and non-respondents are gathered from the Danish Hip Arthroplasty Register.
Sampling Method: Non-Probability Sample
Enrollment: 2777 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Moderate/Severe persistent postsurgical pain | 12-15 months postoperatively
  The main outcome is the number of patients with moderate or severe persistent postsurgical pain in the operated hip, defined as patients with a numerical rating scale (NRS) score higher than 3. The NRS score was dichotomised for the primary outcome because this is more intuitively understood by patients and clinicians. This outcome will be reported as percentage of all patients with 95% confidence interval, which is calculated with assumed binomial distribution as p ± 1.96 √( (p (1 - p) ) / n)

OTHER OUTCOMES:
How satisfied are you with the outcome of your hip replacement surgery? Very satisfied, Satisfied, Neither satisfied nor dissatisfied, Dissatisfied, Very dissatisfied | 12-15 months postoperatively
  Reported as n (%) for each response option. The 1st question assesses overall satisfaction with surgery and have been translated directly from the questionnaire used by the Swedish Arthroplasty Register.
Knowing what your hip replacement surgery did for you, if you could go back in time, would you still have undergone this surgery? Yes, No, Uncertain | 12-15 months postoperatively
  Reported as n (%) for each response option.
Pain frequency: Do you still have pain in the operated hip? Yes, constantly; Yes, daily; Yes, a few times a week; Ja, more rarely; No | 12-15 months postoperatively
  Reported as n (%) for each response option.
Numerical Rating Scale (NRS) pain: Please rate your pain in the operated hip by indicating the number that best describes your pain on average during the last week. 0 means 'No pain' and '10' means 'Pain as bad as you can imagine,' | 12-15 months postoperatively
  Reported as median (interquartile range [IQR]) and number of respondents
Pain domain of the likert-scale version 3.1 of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). | 12-15 months postoperatively
  The five questions in the WOMAC pain domain can be scored 0-4, where 0 is 'none' and 4 is 'extreme'. This results in an overall score of 0-20, which will be reported as median (IQR). Moreover, each response option of the individual questions are reported as n (%).
Pain interference: In total, how much does the pain in the operated hip bother you in your everyday life? Not at all, A little, Some, Much, Very Much | 12-15 months postoperatively
  Reported as n (%) for each response option.
Douleur Neuropathique 4 questions (DN4) interview | 12-15 months postoperatively
  Each of the seven questions in the DN4 interview can be scored 0/1 (no/yes), which results in an overall score of 0-7. A score ≥3 constitutes 'possible' neuropathic pain. Both the median (IQR) DN4 interview score and number of patients (% of all patients) with possible neuropathic pain will be reported.
Other pain: Do you have chronic pain, other than from your operated hip? Yes; No. [If yes] -> Please describe your pain condition: | 12-15 months postoperatively
  Pain conditions will be categorised independently by two authors and reported as n (%).
Analgesic use: Do you take analgesic medication(s) daily or almost daily? Yes; due to pain in the operated hip; Yes, due to other pain; No. [If yes] -> Which medication(s)?: | 12-15 months postoperatively
  Reported as n (%).
Height (cm) | 12-15 months postoperatively
Weight (kg) | 12-15 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Søren Overgaard, MD, PhD, Professor, Study Director — Department of orthopedic surgery, Bispebjerg University Hospital, Denmark
Locations (1):
- Bispebjerg University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
The full dataset will be stored at the Danish national archive (www.rigsarkivet.dk) if possible

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT05845177/Prot_SAP_002.pdf